CLINICAL TRIAL: NCT06930651
Title: A Phase I/II Study of CAR.70-Engineered IL15-Transduced Cord Blood-Derived NK Cells With TGF-beta Receptor 2 (TGFBR2) Knock Out in Conjunction With Lymphodepleting Chemotherapy for the Management of Relapsed/Refractory Myeloid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1967; NCI-2025-02697 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Myeloid Malignancies
MeSH Terms: interventions — Dexamethasone; Cyclophosphamide; fludarabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Escalation with CAR.70 (Experimental): Participants will receive lymphodepleting and primary chemotherapy, followed by a one-time infusion of TGFR KO-CAR27/IL-15 NK cells. Dose of the cells will be a different dose until a maximum tolerated dose is found.
  Interventions: Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Decitabine; Biological: TGFBR2 KO CAR27/IL-15 NK cells
- Phase 2A: Dose Expansion with CAR.70 for AML Patients (Experimental): Participants will receive lymphodepleting and primary chemotherapy, followed by a one-time infusion of TGFR KO-CAR27/IL-15 NK cells using the maximum tolerated dose found in escalation
  Interventions: Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Decitabine; Biological: TGFBR2 KO CAR27/IL-15 NK cells

INTERVENTIONS:
Drug: Dexamethasone — Given Orally
Drug: Cyclophosphamide — Given by IV
Drug: Fludarabine — Given by IV
Drug: Decitabine — Given by IV
Biological: TGFBR2 KO CAR27/IL-15 NK cells — Given by Infusion

SUMMARY:
The goal of this clinical research study is to find the recommended safe dose of TGFBR2 KO CAR27/IL-15 NK cells that can be given to patients with relapsed/refractory disease. The safety and effectiveness of this treatment will also be studied.

DETAILED DESCRIPTION:
This is a phase I/II, two-arm, open-label study. The study will have a phase I dose-escalation portion using a standard "BOIN" approach to determine the MTD of the CAR.70/IL15-transduced/TGFBR2KO CB-NK cells, followed by phase II expansions of 2 arms: 1.) patients with relapsed/refractory AML and 2.) patients with MDS/CMML after HMA failure.

Up to 12 patients will be enrolled in the phase I portion of the study. Following determination of the recommended phase 2 dose (RP2D), 20 patients will be enrolled into the AML arm and 10 patients will be enrolled into the MDS/CMML arm (30 patients total in phase II).

The regimen consists of lymphodepleting and priming chemotherapy with dexamethasone, decitabine, fludarabine and cyclophosphamide, followed by a one-time infusion of the CAR.70/IL15-transduced/TGFBR2KO CB-NK cells

Primary Objectives:

* Phase I: To determine the safety and optimal cell dose of TGFBR2 KO CAR27/IL-15 NK cells in patients with relapsed/refractory myeloid malignances
* Phase II: To determine the response rates of TGFBR2 KO CAR27/IL-15 NK cells in patients with relapsed/refractory AML and in patients with MDS or CMML after HMA failure

Secondary Objectives:

* To determine the CR rate in each cohort
* To determine the rate of flow cytometry MRD negativity (AML cohort only)
* To assess duration of response, relapse-free survival (AML cohort only), and overall survival
* To determine hematologic and non-hematologic toxicities

Exploratory Objectives:

* To assess impact of baseline cytomolecular features and CD70 expression on response
* To quantify persistence of the infused CAR product
* To conduct comprehensive immune reconstitution studies

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Age 18-80 years with diagnosis of:

   1. Relapsed or refractory AML or "treated secondary AML"

      * Patients with a mutation that is targetable with an FDA-approved targeted therapy should have received at least one on these agents. . "Treated secondary AML "includes patients with prior diagnosis of a myeloid neoplasm (e.g. MDS) who received hypomethylating agents for this disease and subsequently progressed to AML. These patients must have received all of the following: a hypomethylating agent + venetoclax and intensive chemotherapy (if a suitable candidate for intensive therapy). These patients may be enrolled at the time of AML diagnosis if they have already received all of the treatments above for their antecedent myeloid neoplasm.
   2. MDS that is intermediate, high-risk or very-high risk by the Revised International Prognostic Scoring System (R-IPSS)

      * Bone marrow blasts must be >5%.
      * The disease must have either 1.) not have responded to at least 4 cycles of a hypomethylating agent or 2.) progressed or relapsed, regardless of the number of cycles received
   3. CMML-1 or CMML-2

      * Bone marrow blasts must be >5%.
      * The disease must have either 1.) not have responded to at least 4 cycles of a hypomethylating agent or 2.) progressed or relapsed, regardless of the number of cycles received
2. CD70 expression >10% measured by immunohistochemistry or multiparameter flow cytometry
3. Performance status </=2 (ECOG Scale)
4. Adequate liver, cardiac, renal and pulmonary function as defined by the following criteria:

   1. Total serum bilirubin </=2 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the PI
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) </=3 x ULN, unless due to the underlying leukemia approved by the PI
   3. Serum creatinine </=2x ULN or creatinine clearance >/=30 mL/min
   4. Left ventricular ejection fraction >/=40% by echocardiogram or MUGA
   5. Oxygen saturation >/=93% on room air
5. Ability to understand and the willingness to sign a written informed consent document
6. Willingness to sign informed consent to long-term follow-up on protocol PA17-0483 to fulfill institutional responsibilities to regulatory agencies
7. Willingness to use adequate contraception prior to study entry, for the duration of study participation, and for 3 months after completion of study participation. For women of childbearing potential, adequate methods of contraception include: complete abstinence,, hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal Ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide.

Exclusion Criteria:

1. Active grade III-V cardiac failure as defined by the New York Heart Association Criteria
2. Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment).
3. Active central nervous system leukemia
4. Known human immunodeficiency virus (HIV) seropositive, unless well-controlled on stable doses of anti-retroviral therapy.
5. Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection Note: Patients who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
6. Patients with a prior or concurrent malignancy whose natural history or treatment is not anticipated to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the PI
7. Use of calcineurin inhibitors (e.g. tacrolimus) within the past 2 weeks
8. Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before lymphodepletion, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator.

   i. Prior recent treatment with corticosteroids, hydroxyurea, and/or cytarabine (up to 2 g/m2 given for cytoreduction within the preceding 7 days) is permitted up until 1 day prior to lymphodepletion.

   • Patients may continue on non-investigational targeted therapies up until 3 days prior to lymphodepletion.
9. Pregnant or breastfeeding women will not be eligible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0
Response rates (AML cohort) | 30 days from CAR infusion
  Rate of complete remission (CR) + CR with incomplete hematologic recovery (CRi) + CR with CR with partial hematologic recovery (CRh)
Response rates (MDS/CMML) cohort | 30 days from CAR infusion
  Rate of CR + partial remission (PR) + CR with limited count recovery (CRL), CRh, hematologic improvement (HI) for MDS; rate of CR + PR + marrow CR (mCR) + clinical benefit (CB) for CMML

SECONDARY OUTCOMES:
CR rate | 30 days from CAR infusion
  Rate of CR in each cohort
Measurable residual disease (MRD) negativity (AML cohort) | 30 days from CAR infusion
  Rate of MRD negativity assessed by flow cytometry
Duration of response | Through study completion; an average of 1 year
  Time from response to relapse
Relapse-free survival | Through study completion; an average of 1 year
  Time from response to relapse or death from any cause
Overall survival | Through study completion; an average of 1 year
  Time from treatment start to death from any cause
Hematologic and non-hematologic toxicities | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org